CLINICAL TRIAL: NCT06444958
Title: Morbidity and Mortality Rates Among Children Aged 0-59 Months: A Cross-sectional Study From Mogadishu, Somalia
Brief Title: Morbidity and Mortality Rates Among Children Aged 0-59 Months
Status: Completed | Type: Observational
Sponsor: Kalkaal Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KHRC2024/050
Record Dates: First submitted 2024-05-30; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Morbidity;Infant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: observational study without any intervention component. — extracting and analyzing the following data:
  Outpatient department records: Diagnoses, treatments, patient demographics Inpatient admission records: Admission diagnoses, treatments, patient outcomes (discharged, transferred, died) Mortality records: Causes of death for pediatric patients

SUMMARY:
This retrospective observational study aimed to investigate the patterns of morbidity and mortality among children under 5 years of age in the population served by Kalkaal Hospital. Researchers analyzed 2023 data from the hospital's electronic medical records and administrative databases to identify the most common pediatric diagnoses and causes of illness and death in this community.

DETAILED DESCRIPTION:
This study investigated the patterns of morbidity and mortality among children under 5 years of age in the population served by Kalkaal Hospital. The specific objectives were to:

Identify the most common diagnoses and causes of illness and death in the under-5 population presenting to Kalkaal Hospital.

Analyze demographic factors (e.g. age, sex) associated with certain disease profiles and health outcomes.

Evaluate treatment practices, health service utilization, and mortality rates for the key pediatric health issues identified.

Provide a comprehensive epidemiological assessment of the burden of childhood illness and mortality in this local community.

Methods:

This was a retrospective, observational study that analyzed 2023 data from the electronic medical records and administrative databases of Kalkaal Hospital. The researchers extracted and analyzed the following data:

Outpatient department records: Diagnoses, treatments, patient demographics Inpatient admission records: Admission diagnoses, treatments, patient outcomes (discharged, transferred, died) Mortality records: Causes of death for pediatric patients The data was cleaned, coded, and analyzed using statistical software. Descriptive statistics were calculated to characterize the morbidity and mortality patterns. Regression analyses were conducted to identify demographic and clinical factors associated with key health outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 0-59 months who were admitted to Kalkaal Hospital during the specified study period.
2. Medical records with complete and adequate information regarding age, gender, presenting symptoms, and diagnoses.

   -

Exclusion Criteria:

1. Children outside the age range of 0-59 months.
2. Medical records with missing or incomplete information necessary for the analysis.
3. Children admitted to Kalkaal Hospital for reasons unrelated to the study objectives (adult patients, non-pediatric cases).

Ages: 0 Months to 59 Months | Sex: All
Age Groups: Child
Study Population: Children under 5 years of age in the population served by Kalkaal Hospital
  The target population was the pediatric patients under the age of 5 who accessed healthcare services at Kalkaal Hospital.
  The researchers extracted data from the hospital's records on all children under 5 who presented as outpatients, were admitted as inpatients, or were recorded in the mortality database.
Sampling Method: Probability Sample
Enrollment: 1675 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Morbidities: Incidence rates of various morbidities among children presenting to the outpatient department and inpatient wards. | JANUARY-DECEMBER 2023
  This outcome measure will calculate the incidence rates of various morbidities among children under 18 years of age who presented to the Kalkaal Hospital outpatient department or were admitted to the inpatient wards during the 5-year study period (2018-2022). The incidence rates will be reported for the top 10 most common morbidities observed in the study population.
Mortality Rate by Age Group: Mortality rates and associated risk factors across different age groups of children under 18 (under 28 days, 29-365 days, 1-5 years). | JANUARY-DECEMBER 2023
  This outcome measure will determine the mortality rates among children under 18 years of age treated at Kalkaal Hospital, stratified by the following age groups: under 28 days, 29-365 days, and 1-5 years. The analysis will also identify risk factors associated with mortality in each age group.
Average Length of Hospital Stay: Median hospital stay duration for children under 18 years old. | JANUARY-DECEMBER 2023
  This outcome measure will calculate the median length of hospital stay for children under 18 years old who were admitted to the Kalkaal Hospital inpatient wards during the study period. The average length of stay will be reported overall, as well as by primary diagnosis categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Kalkaal Hospital, Mogadishu, Banadir, Somalia

IPD SHARING:
Plan to Share IPD: Undecided
Data Sharing Plan:
  The de-identified individual patient data (IPD) collected and analyzed for this retrospective observational study on pediatric morbidity and mortality at Kalkaal Hospital will be made available to other researchers upon reasonable request.